Accuracy of dental implant placement using dynamic navigation or the freehand method: a randomized controlled clinical trial in novice operators

Document date: August 30, 2023

## Faculty of Medicine and Health Sciences Bellvitge, L'Hospitalet de Llobregat





## INFORMED CONSENT

Accuracy of dental implant placement using dynamic navigation or the freehand method: a randomized controlled clinical trial in novice operators

I, ... (patient's full name)...., of legal age, with DNI ... (patient's full DNI)...., acting in my own name and interest, freely accept to participate in the research: "Accuracy of dental implant placement using dynamic navigation or the freehand method: a randomized controlled clinical trial in novice operators".

## I declare that

I have received information about the project, I have understood its meaning and objectives.

I have read the information sheet given to me.

I have been able to ask questions about the study.

I have received sufficient information about the study.

I have spoken to: .....

(name of investigator)

-I understand that my participation is voluntary and that the data will be collected under the conditions detailed in the Patient Information Sheet.

According to the General Data Protection Regulation, consent to the processing of your personal data and to their transfer is revocable. You may exercise your right of access, rectification and cancellation by contacting the researcher.

- I understand that I can withdraw from the study:
  - Whenever I want.
  - Without having to explain myself.
  - Without affecting my medical care.

I freely give my consent to participate in the study "Accuracy of dental implant placement using dynamic navigation or the freehand method: a randomized controlled clinical trial in novice operators" and I allow the principal investigator (Victor Ruiz Romero) and his research team to manage my personal data and to keep all the records made about me, with the guarantees and the legally foreseen deadlines.

Signature of Patient Signature of Investigator

Name: Name:

Date:

Date: